CLINICAL TRIAL: NCT06092385
Title: SASL Swiss Cirrhosis Cohort Study
Brief Title: SASL Swiss Cirrhosis Cohort
Acronym: SSCiCoS
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-01370; bb23Bernsmeier
Record Dates: First submitted 2023-10-09; First posted 2023-10-23 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Liver Cirrhosis
Keywords: SASL Swiss Cirrhosis Cohort Study (SSciCoS); chronic liver disease
MeSH Terms: conditions — Liver Cirrhosis | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum and plasma. Other biological material (e.g. ascites, urine, liver biopsies, liver resections, gut biopsies), sampled routinely for clinical reasons: stored for research purpose. Excess tissue will only be used for research purposes when the histopathology department has performed a full evaluation and no further tissue would be required for clinical diagnostic purposes. Liver or gut tissue will be used immediately, formalin-fixed and paraffin-embedded or snap-frozen and stored at -80°C. Also archived previously sampled tissue might be investigated in retrospect upon recruitment into the study. If possible, white blood cells from fluids (ascites, urine) will be separated by density centrifugation and either used immediately or stored at -140°C. The fluid supernatant will also be collected and stored at -80°C in de-centralised biobanking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with chronic liver disease and histologically proven cirrhosis
  Interventions: Other: Data collection
- Control subjects with no signs of cirrhosis
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Clinical assessment and blood sampling at day of inclusion and in 6- monthly intervals for stable cirrhotic patients; at day of inclusion and on days 3, 7, 14 and 28 for acute decompensation or acute-on-chronic liver failure patients; assessment of clinical, psychosocial/behavioural and patient-reported data in parallel with blood sampling;
  * Biobanking of PBMCs and serum/plasma samples
  * Biobanking of other biological material if sampled for clinical reasons (liver biopsies, ascites, urine, gut mucosa, lymph nodes)

SUMMARY:
This is a national prospective long-term multicentre observational cohort study following patients with cirrhosis in order to systematically and longitudinally record epidemiological, clinical, histological, psychosocial and patient-reported data and biobank biological material from patients with cirrhosis.

The central element of all scientific operation and productivity in the Swiss Cirrhosis Cohort Study (SSCiCoS) is the so-called "nested project" (NP). Based on the evolving large pool of data and biological samples, SSCiCoS investigators use the data pool in order to investigate specific hypotheses and questions.

DETAILED DESCRIPTION:
For patients with end-stage cirrhosis there are no treatment options other than transplantation, a medically and ethically challenging procedure. The challenge therefore is to prevent the need for liver transplantation in as many patients with cirrhosis as possible.

In order to reach this aim, patients with cirrhosis should be identified and followed regularly according to the highest standard of current knowledge. Numerous aspects of the disease need to be detailed: its epidemiology in Switzerland, its pathophysiology including the mechanism of scar tissue generation and resolution, the associated immune dysfunction and subsequent organ failures, disease related psychosocial and behavioural factors, perceived burden of liver cirrhosis in patients, diagnostic and prognostic biomarkers for disease dynamics, both progression and regression of disease, and stage-specific therapeutic strategies.

This is a national prospective long-term multicentre observational cohort study following patients with cirrhosis in order to systematically and longitudinally record epidemiological, clinical, histological, psychosocial and patient-reported data and biobank biological material from patients with cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* A) Patients with chronic liver disease and histologically proven cirrhosis
* B) Control subjects with no signs of cirrhosis

Exclusion Criteria:

* Age <18 years
* patients who developed hepatocellular carcinoma (HCC) and/or cholangiocellular carcinoma (CCC)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The SSCiCoS enrols patients with chronic liver disease and histologically proven cirrhosis presenting at any of the participating centres. Additionally control subjects will be included who do not have evidence for the presence of cirrhosis. These control subjects may involve healthy controls as well as patients (pathological controls). In theory any adult subject with no suscpicion of cirrhosis, HCC or CCC may be included. The concomittent built-up of the control cohort is supposed to serve as control for the cirrhosis patients involved, thus specifically, but not exclusively healthy age-matched controls as well as pathological controls presenting with a pathology or events similar to the condition and/or complications of cirrhosis (e.g. chronic liver disease with no cirrhosis, non-cirrhotic portal hypertension, ascites, infection, gastrointestinal bleeding or acute kidney injury of other origin than cirrhosis).
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2024-06-04 (Actual); Primary Completion 2033-01 (Estimated); Study Completion 2033-01 (Estimated)

PRIMARY OUTCOMES:
Change in Number of liver transplantations | Through study completion, an average of 10 years
  Change in Number of liver transplantations
Change in Number of survival | Through study completion, an average of 10 years
  Change in Number of survival
Change in Number of transplant free survival | Through study completion, an average of 10 years
  Change in Number of transplant free survival
Change in Number of decompensation events | Through study completion, an average of 10 years
  Change in Number of decompensation events
Change in Number of organ failure | Through study completion, an average of 10 years
  Change in Number of organ failure
Change in Number of infectious complications | Through study completion, an average of 10 years
  Change in Number of infectious complications
Change in Number of maligancies | Through study completion, an average of 10 years
  Change in Number of maligancies
Change in Patient Reported Outcome Measures (PROMs, e.g. Epworth Sleepiness Scale) | Through study completion, an average of 10 years
  The Epworth Sleepiness Scale is a subjective measure of a patient's sleepiness. The test is a list of eight situations in which the tendency to become sleepy on a scale of 0 (no chance of dozing) to 3 (high chance of dozing) is rated. (0 - 10: Normal range; 10 - 12: Borderline; 12 - 24: Abnormal)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Bernsmeier, Prof. Dr. med., Principal Investigator — University Centre for Gastrointestinal and Liver Diseases, University Hospital Basel, Switzerland
Locations (10):
- Switzerland (10):
  - Gastroenterology and Hepatology, Cantonal Hospital Ticino, Lugano, Canton Ticino
  - University Centre for Gastrointestinal and Liver Diseases, University Hospital Basel, Switzerland, Basel
  - Department of Visceral Surgery and Medicine, University Hospital of Berne, Bern
  - Gastroenterology and Hepatology, University Hospital Geneva, Geneva
  - Gastroenterology and Hepatology, Lausanne University Hospital, Lausanne
  - Ticino Liver Centre, Lugano
  - Gastroenterology and Hepatology, Cantonal Hospital St. Gallen, Sankt Gallen
  - Arud Centre for addiction medicine Zurich, Zurich
  - Digestive Diseases Insti- tute GastroZentrum, Hirslanden Clinic Zurich, Zurich
  - Gastroenterology and Hepatology, University Hospital Zurich, Zurich